CLINICAL TRIAL: NCT02367651
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study of Pazopanib Versus Placebo as Maintenance Therapy for Patients Who Have Not Progressed After First-line Chemotherapy for Advanced Soft Tissue Sarcoma (STS)
Brief Title: Study of Pazopanib Versus Placebo as Maintenance Therapy for Advanced Soft Tissue Sarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study cancelled: Withdrawn before enrollment of any participants
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201187
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Soft tissue sarcoma; Pazopanib; Tyrosine kinase inhibitor
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pazopanib (Experimental): Subjects will receive pazopanib 800 mg once daily during each 28-day treatment period until disease progression, unacceptable adverse event (AE)/serious adverse event (SAE), death or withdrawal of consent
  Interventions: Drug: Pazopanib 800 mg
- Placebo (Placebo Comparator): Subjects will receive placebo once daily during each 28-day treatment period until disease progression, unacceptable AE/SAE, death or withdrawal of consent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pazopanib 800 mg — Aqueous film-coated, oval-shaped, white tablets containing either 200 mg or 400 mg pazopanib
  Arms: Pazopanib
Drug: Placebo — Tablets matching the 200 mg and 400 mg pazopanib tablets
  Arms: Placebo

SUMMARY:
Pazopanib monotherapy is approved by the Food and Drug Administration (FDA), European Medicines Agency, and other regulatory authorities worldwide for the treatment of patients with advanced renal cell carcinoma and patients with advanced soft tissue sarcoma (STS) who received prior chemotherapy. Based on the improved progression-free survival and sustained responses observed in a pivotal Phase 3, randomized, placebo-controlled study, it is hypothesized that pazopanib may have a role in a maintenance setting for STS in maintaining the initial response to chemotherapy and delaying the need for further treatment at relapse and its associated toxicity and impact on health-related quality-of-life. This Phase 2, randomized, double-blind, placebo-controlled study will evaluate maintenance therapy with pazopanib versus placebo in subjects with advanced or metastatic STS who have not progressed after 4 to 6 cycles of first-line anthracycline-based chemotherapy. Approximately 188 eligible subjects will be randomized in a 1:1 ratio to treatment with pazopanib 800 milligrams (mg) daily or placebo. Study completion will be the point at which 70% of randomized subjects have died. Once a subject has objective evidence of disease progression, the subject will be managed as per standard practice by their physician. Subjects will continue to be followed for second progression, health related quality of life, survival until study completion, withdrawal of consent, or early termination of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent before performing study-specific procedures or assessments and are willing to comply with treatment and follow-up.
* Age >= 18 years
* Have a local histopathological diagnosis of one the following STS tumor types based on World Health Organization (WHO) 2013 classification. Fibroblastic (adult fibrosarcoma, myxofibrosarcoma, sclerosing epithelioid fibrosarcoma, malignant solitary fibrous tumors), Leiomyosarcoma , Vascular (epithelioid haemangioendothelioma, angiosarcoma), Skeletal muscle (pleomorphic and alveolar rhabdomyosarcoma only), Malignant peripheral nerve sheath tumors, Malignant glomus tumors, Alveolar soft part sarcoma, Uncertain differentiation (synovial, epithelioid, clear cell, desmoplastic small round cell, extra-renal rhabdoid, malignant mesenchymoma, perivascular epithelioid cell tumor [PEComa], intimal sarcoma), Undifferentiated soft tissue sarcomas (undifferentiated pleomorphic sarcoma or undifferentiated not otherwise specified), Other types of sarcoma not in listed exclusion criteria (contact medical monitor in case of unclear eligibility of a given subtype)
* Completed 4 to 6 cycles of first-line anthracycline-based chemotherapy for metastatic disease without disease progression.

Note: Subjects must have no evidence of radiological progression as confirmed by Computed Tomography (CT)/ Magnetic Resonance Imaging (MRI) within 4 weeks before randomization and no signs of clinical progression before randomization.

* The date of study randomization must be 3 to 8 weeks following the last dose of chemotherapy. All chemotherapy-related side effects (except alopecia) must have resolved to grade 1 or better.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Able to swallow and retain oral tablets.
* Adequate baseline organ function
* Baseline Left Ventricular Ejection Fraction (LVEF) above lower limit of normal (LLN) based on institution's normal range.
* Corrected QT interval (QTc) <450 milliseconds (msec) or QTc <480 msec for subjects with bundle branch block. For subject eligibility and withdrawal, Bazett's QT correction formula (QTcB) will be used. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of the first dose of study treatment and agree to use effective contraception, as defined in Study Protocol during the study and for 14 days following the last dose of study treatment.

Note: Female subjects who are lactating must discontinue nursing before the first dose of study treatment and refrain from nursing from the first dose until 14 days following the last dose of study treatment.

* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Prior malignancy. Note: Subjects who have had another malignancy and have been disease-free for 3 years or more, or subjects with a history of completely resected non-melanoma skin carcinoma or successfully treated in situ carcinoma are eligible.
* Any of the following tumor types: Adipocytic sarcoma (all subtypes) , All rhabdomyosarcoma that are NOT alveolar or pleomorphic, Chondrosarcoma, Osteosarcoma, Ewing tumors / primitive neuroectodermal tumor (PNET), Gastro-intestinal stromal tumors (GIST), Dermofibromatosis sarcoma protuberans, Inflammatory myofibroblastic sarcoma, Malignant mesothelioma, Mixed mesodermal tumors of the uterus (carcinosarcoma), Subjects with low grade histology (French Fédération Nationale des Centres de Lutte Contre le Cancer [FNCLCC] grade 1 or those with incomplete grading information FNCLCC grade X)
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding within 28 days before beginning study treatment.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to: Malabsorption syndrome, Major resection of the stomach or small bowel
* History of any one or more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting, Myocardial infarction, Unstable angina, Coronary artery bypass graft surgery, Symptomatic peripheral vascular disease, Class III or IV congestive heart failure (CHF), as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension (defined as systolic blood pressure [SBP] >=140 millimeters of mercury (mmHg) or diastolic blood pressure [DBP] >= 90 mmHg)
* History of cerebrovascular accident (CVA), transient ischemic attack (TIA), pulmonary embolism (PE), or deep venous thrombosis (DVT) within the past 6 months unless therapeutically coagulated for at least 6 weeks.
* Major surgery or trauma within 28 days before the first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.

Note: Lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching but not infiltrating (abutting) the vessel is acceptable (CT with contrast is strongly recommended to evaluate such lesions).

* Recent hemoptysis (>= 1/2 teaspoon or 2.5 milliliters of red blood) within 8 weeks of the first dose of study drug.
* Any of the following hepatic or biliary conditions:

Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months before the first dose of study treatment. Exception: subject can be enrolled if hepatitis C Ribonucleic acid (RNA) is negative.

Presence of another active liver or biliary disease. Exceptions: subject can be enrolled in case of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment.

Note: Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, persistent jaundice, or cirrhosis.

* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* A positive pre-study alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or 5 half-lives of a drug (whichever is longer) before the first dose of study treatment and for the duration of the study.
* Treatment with any of the following anti-cancer therapies: Radiation therapy, surgery or tumor embolization within 14 days before the first dose or pazopanib OR chemotherapy, immunotherapy, biologic therapy (including prior pazopanib or other Vascular Endothelial Growth Factor (VEGF), Platelet-Derived Growth Factor Receptor [PDGFR], or Cytokine Receptor [c-Kit] inhibitor), investigational therapy, or hormonal therapy within 14 days or 5 half-lives of a drug (whichever is longer) before the first dose of pazopanib.
* A known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or excipients that contraindicate their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | At Day 57 and every 8 weeks thereafter until disease progression or death (assessed up to 2 years)
  PFS is defined as time from randomization to development of disease progression or death due to any cause. Disease progression will be evaluated based on investigators' radiologic assessments by Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | At Day 57, then every 8 weeks until disease progression, and every 3 months thereafter until death (assessed up to 2 years)
  OS is defined as time from randomization to death due to any cause.
Disease control rate (DCR) | At 4 months after randomization
  DCR is defined as percentage of complete response + partial response + stable disease at 4 months after randomization based on RECIST version 1.1.
Safety and tolerability as assessed by physical examination findings | From Day 1 up to end of treatment (assessed up to 2 years)
  A brief physical examination will include height (baseline only), body weight and evaluation of the subject's medical conditions
Safety and tolerability as assessed by temperature measurement | From Day 1 up to end of treatment (assessed up to 2 years)
Safety and tolerability as assessed by systolic and diastolic blood pressure measurement | From Day 1 up to end of treatment (assessed up to 2 years)
Safety and tolerability as assessed by pulse rate measurement | From Day 1 up to end of treatment (assessed up to 2 years)
Safety and tolerability as assessed by composite of clinical laboratory tests | From Day 1 up to end of treatment (assessed up to 2 years)
  Clinical laboratory tests will include chemistry and hematology parameters
Safety and tolerability as assessed by cardiac assessments | From Day 1 up to end of treatment (assessed up to 2 years)
  Cardiac assessments will include twelve-lead electrocardiogram (ECG), echocardiogram (ECHO) or multigated angiogram (MUGA) assessments
Safety and tolerability as assessed by number of subjects with adverse event | From Day 1 up to end of treatment (assessed up to 2 years)
Time to worsening of dyspnea or pain scores as measured by the MD Anderson Symptom Inventory (MDASI) questionnaire | Weekly from baseline up to week 48
  The MDASI is a 19-item general cancer questionnaire asking subjects to rate symptoms at their worst on a scale of 0-10, including pain and shortness of breath as items. Time to symptom deterioration is defined as worsening in tumour pain score or dyspnea score of 2 points or more from baseline, confirmed by at least one additional weekly measure within a four week period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline